CLINICAL TRIAL: NCT05787431
Title: Levels of Physical Activity After SARS-CoV-2 Infection in Greek Adults: the Role of Pre-illness Vaccination and the Number of Reinfections.
Brief Title: Levels of Physical Activity After SARS-CoV-2 Infection in Pre-illness Vaccinated and Unvaccinated Greek Adults.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emmanouil D. Zacharakis (Other)
Responsible Party: Sponsor-Investigator, Emmanouil D. Zacharakis, Emmanouil D. Zacharakis, emzach@phed.uoa.gr, +306977915982, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Other Study IDs: 1454/11-01-2023
Record Dates: First submitted 2023-03-21; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 (Coronavirus Disease 2019)
Keywords: Physical Activity, exercise, public health, Post COVID
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unvaccinated individuals: COVID-19 recovered individuals who are not been vaccinated with any dose of COVID-19 vaccines.
- Vaccinated individuals: COVID-19 recovered individuals who are vaccinated with one or more dose of COVID-19 vaccines, and stratified by sub-groups.

SUMMARY:
Coronavirus infection has an impact on several aspects of everyday life including the levels of Physical Activity (PA). Investigators wish to (1) detect changes on PA levels in recovered SARS-CoV-2 (COVID-19) adults compared to the pre-infection levels and (2) identify a potential relationship between changes of PA levels and pre-illness vaccination profile along with individual's number of infection/reinfections. It is assumed that the impact of COVID-19 infection on PA would be more pronounced in cases of repeated infections and/or in the unvaccinated compared to the vaccinated individuals against COVID-19.

DETAILED DESCRIPTION:
Coronavirus identified in 2019, SARS-CoV-2 (COVID-19), has caused a pandemic of respiratory illness in which manifestation ranging from asymptomatic presentation to critically illness with severe pneumonia, acute respiratory distress syndrome, respiratory failure, or multiple organ failure. It may influence several aspects of everyday life including the levels of Physical Activity such as walking, cycling, sports or active recreation and, thus, has negative effect on general health and quality of life. Recent findings demonstrate a relation between COVID-19 infection and impairment in functional capacity, and suggest that may also be associated with an increased risk of acute and post-acute death. Moreover, individuals who have been infected might suffer long-term consequences as a result of their infection (Long COVID), for few weeks (short term) or 10-20 weeks (medium term) or more than six months (long term) post-infection.

The current study is designed to assess changes in PA (overall and in four domains i.e. daily occupation, transportation to and from daily occupation, leisure time activities, and regular sporting activities) caused by COVID-19 infection (i.e. in the short term, 4 weeks post infection) concerning the pre-illness vaccination profile and the number of infections/reinfections using a web-based validated questionnaire in a large population of Greece. Investigators hypothesize that the impact of COVID-19 infection on PA levels would be more pronounced in cases of repeated infections and/or in the unvaccinated compared to the vaccinated individuals against COVID-19. With regard to the potential burden of COVID-19 in functional capacity, investigators wish:

1. to detect changes on PA levels in recovered COVID-19 adults compared to the pre-infection levels as a result of a post-effect impact;
2. to identify a potential relationship between changes of PA levels and pre-illness vaccination profile along with individual's number of infection/reinfections so as to detect correlations amongst different parameters.

The Greek version of the revised Active-Q (AQGR) which is a self-reported, online, interactive physical activity questionnaire that assesses adult's habitual activity on weekly basis (in four main PA domains: daily occupation, transportation to and from daily occupation, leisure time activities, and regular sporting activities) is employed. Regarding questions of medical treatment during COVID-19 infection, individual's number of infection/reinfections and other relative parameters, additional questionnaire items have been incorporated. In total, the current web-based questionnaire consisted of 60-67 questions, based on previous responses and follow-up patterns, and will be extensively used to address the aims of the current study.

ELIGIBILITY:
Inclusion Criteria:

COVID-19 recovered individuals aged from 18 to 80 years old.

Exclusion Criteria:

Individuals without any confirmed COVID-19 infection, severe musculoskeletal problems, cognitive impairment/dementia, participation in any strict weight loss control program, gestation or childbirth within one year of the study's start date.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 recovered individuals aged from 18 to 80 years old who are residents of Greece and have been diagnostically confirmed with COVID-19 infection and recovered at least one month before answering the survey instrument.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Levels of Physical Activity (PA) | One (1) month at least after recovery from COVID-19 infection
  Levels of PA, before and after COVID-19 infection, will be recorded

OTHER OUTCOMES:
Protective effect of vaccination in post-COVID-19 burden on Physical Activity (PA) | One (1) month at least after recovery from COVID-19 infection
  Correlations between the number of doses of vaccines and the post-COVID-19 burden on PA will be performed
The role of the number of re-infections and post-COVID-19 burden on PA | One (1) month at least after recovery from the last COVID-19 infection
  Correlations between the number of re-infections and the post-COVID-19 burden on PA will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil D. Zacharakis, PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- National and Kapodistrian University of Athens, Athens, Attica, Greece

REFERENCES:
- [Result] Bourdas DI, Zacharakis ED. Impact of COVID-19 Lockdown on Physical Activity in a Sample of Greek Adults. Sports (Basel). 2020 Oct 21;8(10):139. doi: 10.3390/sports8100139. PMID 33096721
- [Result] Bourdas DI, Zacharakis ED, Travlos AK, Souglis A, Georgali TI, Gofas DC, Ktistakis IE, Deltsidou A. Impact of lockdown on smoking and sleeping in the early COVID-19 presence: Datasets of Greek Adults sample. Data Brief. 2021 Dec;39:107480. doi: 10.1016/j.dib.2021.107480. Epub 2021 Oct 14. PMID 34664028
- [Result] Bourdas DI, Zacharakis ED. Evolution of changes in physical activity over lockdown time: Physical activity datasets of four independent adult sample groups corresponding to each of the last four of the six COVID-19 lockdown weeks in Greece. Data Brief. 2020 Oct;32:106301. doi: 10.1016/j.dib.2020.106301. Epub 2020 Sep 11. PMID 32934972
- [Result] Bourdas DI, Zacharakis ED, Travlos AK, Souglis A. Return to Basketball Play Following COVID-19 Lockdown. Sports (Basel). 2021 Jun 3;9(6):81. doi: 10.3390/sports9060081. PMID 34204988
- See also: Official web-page of the study — https://hub.uoa.gr/the-impact-of-the-disease-and-re-infections-of-covid-19-on-physical-activity-in-a-vaccinated-and-non-vaccinated-population-in-greece/